CLINICAL TRIAL: NCT07192835
Title: Effect of Fruit Elicitation With Melatonin on Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Vicente Agulló García, Doctor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DTA.VAG.240905
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Dietary Bioavailability; Plant Extracts; Phenolic Compounds; Melatonin
Keywords: Melatonin; Phenolic compounds; Flavanones; Anthocyanins; Lemon; Blood orange; Sweet cherry; Bioavailability; Human Nutrition; Functional Foods; Sustainable Agriculture

STUDY DESIGN:
Intervention Model Description: This is a randomized, acute, crossover study. Each participant will consume juice from both melatonin-treated fruits and untreated fruits in different periods, with a 15-day washout interval between interventions. All participants act as their own control, allowing direct comparison of bioactive compound absorption and metabolism between treated and untreated fruits. The order of interventions will be randomized to minimize sequence effects.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin-treated fruit first, then control fruit (Experimental): Participants will consume juice prepared from melatonin-treated fruits (lemon, blood orange, or sweet cherry) during the first intervention period, followed by juice from untreated control fruits after a 15-day washout period. Urine samples will be collected at specified intervals to measure bioactive compound absorption and metabolism.
  Interventions: Dietary Supplement: Juice from untreated control fruits; Dietary Supplement: Juice from melatonin-treated fruits
- Control fruit first, then melatonin-treated fruit (Experimental): Participants will consume juice prepared from untreated control fruits (lemon, blood orange, or sweet cherry) during the first intervention period, followed by juice from melatonin-treated fruits after a 15-day washout period. Urine samples will be collected at specified intervals to measure bioactive compound absorption and metabolism.
  Interventions: Dietary Supplement: Juice from untreated control fruits; Dietary Supplement: Juice from melatonin-treated fruits

INTERVENTIONS:
Dietary Supplement: Juice from untreated control fruits — Participants will consume 300 g of juice prepared from untreated fruits (lemon, blood orange, or sweet cherry) under fasting conditions on the intervention day. Urine samples will be collected at 0-3.5 h, 3.5-12 h, and 12-24 h post-consumption to assess absorption and metabolism of bioactive compounds.
Dietary Supplement: Juice from melatonin-treated fruits — Participants will consume 300 g of juice prepared from fruits (lemon, blood orange, or sweet cherry) treated preharvest with melatonin (0.1, 0.3, or 0.5 mM). Juice will be consumed under fasting conditions on the intervention day. Urine samples will be collected at 0-3.5 h, 3.5-12 h, and 12-24 h post-consumption to assess absorption and metabolism of bioactive compounds.

SUMMARY:
The goal of this clinical trial is to learn if treating fruits with melatonin helps the body absorb and use healthy plant compounds. It will also learn how much melatonin from the fruits is taken up by the body. The main questions it aims to answer are:

* Does melatonin treatment of fruits raise the amount of healthy compounds the body absorbs?
* Does melatonin from treated fruits appear in urine after eating them?

Researchers will compare juice made from melatonin-treated fruits to juice made from untreated fruits to see if melatonin changes absorption.

Participants will:

* Follow a special low-plant-compound diet for 3 days before each test day
* Drink 300 grams of juice from treated or untreated fruit while fasting
* Provide urine samples before and after drinking the juice
* Return 15 days later to switch to the other juice type
* Repeat this process with lemon, blood orange, and cherry

DETAILED DESCRIPTION:
This clinical trial will investigate whether melatonin treatments in fruits can improve the bioavailability of bioactive compounds in humans. Melatonin is a natural molecule with antioxidant and protective properties. Its preharvest application has been shown to enhance postharvest fruit quality and raise the levels of phenolic compounds such as flavanones and anthocyanins. However, it is not yet known whether these changes in fruit composition result in greater absorption and metabolism of these compounds in humans after fruit consumption. The central hypothesis is that melatonin-treated fruits will show increased concentrations of bioactive compounds and melatonin, leading to higher bioavailability and urinary excretion of these compounds and their metabolites compared to untreated fruits. This would provide evidence that a sustainable agronomic practice can enhance not only fruit quality but also its nutritional and functional value for human health.

The study will follow a randomized acute crossover design with 20 healthy adult participants. Volunteers will consume juices prepared from melatonin-treated or untreated lemons, blood oranges, and sweet cherries under fasting conditions. Each participant will act as their own control, with a washout period of 15 days between interventions. To reduce variability, participants will follow a controlled low-phenolic and low-melatonin diet for three days before each test day. On the intervention day, urine samples will be collected before juice intake and at several time intervals over the following 24 hours (0-3.5 h, 3.5-12 h, and 12-24 h). Samples will be analyzed to determine the excretion of phenolic compounds, melatonin, and their metabolites, normalized by total urine volume. Fruits will be characterized using ultra-high-performance liquid chromatography coupled with triple quadrupole mass spectrometry (UHPLC-QqQ-MS/MS), and the same methodology will be applied to urine samples to provide precise and reliable quantification.

This project is of high scientific, social, and economic interest. From a scientific perspective, it will generate new knowledge about the bioavailability of bioactive compounds from melatonin-treated fruits, addressing a current gap in the understanding of how preharvest treatments influence not only fruit quality but also the absorption and metabolism of phenolics and melatonin in humans. These results may open new research avenues on the impact of sustainable agricultural strategies on human nutrition and health. From a social perspective, the study is aligned with increasing concerns about metabolic and cardiovascular diseases and with consumer demand for healthier foods. Understanding how to optimize the bioavailability of beneficial compounds through preharvest practices could promote dietary patterns that support better health. From an economic perspective, the trial focuses on fruits with Protected Geographical Indication (PGI), such as Valencian citrus and Alicante cherries. Demonstrating added nutritional and functional value through melatonin treatments could raise the competitiveness and market appeal of these products, supporting producers and the agro-food sector.

The feasibility of the study is guaranteed by access to the necessary resources and infrastructure. The fruits will be sourced from PGI-certified orchards in the Valencian Community, cultivated under conventional practices, and harvested at commercial maturity to ensure optimal quality. Melatonin treatments will be applied using manual sprayers at key stages of fruit development. The human intervention will take place at the Miguel Hernández University (UMH), where facilities are available to conduct the study and handle biological samples. Urine will be collected and stored at -80 °C until analysis to preserve sample integrity. The analytical laboratory is fully equipped with UHPLC and tandem mass spectrometry systems and has validated protocols for phenolic and melatonin analysis, developed in previous studies by the research team. The investigators have extensive experience in plant bioactives, fruit physiology, and human nutrition, ensuring proper execution of the project.

In summary, this study is innovative, multidisciplinary, and highly feasible. It will provide important insights at the intersection of agriculture, food science, and human health, with potential benefits for society, the scientific community, and the agro-food industry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-65 years
* Body mass index (BMI) between 18.5 and 24.9 kg/m²
* Non-smokers
* No chronic diseases (such as diabetes, cardiovascular disease, or cancer)
* Not taking regular medication
* Willing to follow a diet low in phenolic compounds and melatonin during the study periods
* Able and willing to provide urine samples according to study instructions

Exclusion Criteria:

* Presence of chronic diseases or metabolic disorders
* Use of medications that could affect metabolism or absorption of compounds
* Smoking or use of nicotine products
* Allergies or intolerance to citrus fruits or cherries
* Pregnancy or breastfeeding
* Inability or unwillingness to comply with study procedures or dietary restrictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Biodisponibility of phenolic compounds and melatonin from melatonin-treated fruits | 0-3.5, 3.5-12, and 12-24 hours post-consumption for each intervention period
  The primary outcome is the amount of phenolic compounds (flavanones and anthocyanins) and melatonin absorbed and excreted by participants after consuming 300 g of juice from melatonin-treated fruits. Urine samples are collected at 0-3.5 h, 3.5-12 h, and 12-24 h post-consumption, and concentrations are measured using UHPLC-QqQ-MS/MS. Excretion is normalized to creatinine to account for urine volume differences.

CONTACTS AND LOCATIONS:
Locations (1):
- University Miguel Hernandez, Orihuela, Alicante/Alacant, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agullo V, Villano D, Garcia-Viguera C, Dominguez-Perles R. Anthocyanin Metabolites in Human Urine after the Intake of New Functional Beverages. Molecules. 2020 Jan 16;25(2):371. doi: 10.3390/molecules25020371. PMID 31963236
- [Background] Agullo V, Dominguez-Perles R, Moreno DA, Zafrilla P, Garcia-Viguera C. Alternative Sweeteners Modify the Urinary Excretion of Flavanones Metabolites Ingested through a New Maqui-Berry Beverage. Foods. 2020 Jan 3;9(1):41. doi: 10.3390/foods9010041. PMID 31947712